CLINICAL TRIAL: NCT05647941
Title: Non-invasive Response Assessment of Neo-adjuvant Chemotherapy in Gastric Cancer Patients Based on Circulating Exosomal LncRNA-GC1
Brief Title: Neo-adjuvant Chemotherapy Evluation in Gastric Cancer Patients Based on Circulating Exosomal LncRNA-GC1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, Director of Department of General Surgery, Chinese PLA General Hospital, Chinese PLA General Hospital
Other Study IDs: neo-Biomarker
Record Dates: First submitted 2022-12-04; First posted 2022-12-13 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Gastric Cancer; Chemotherapy Effect
Keywords: Circulating exosomal lncRNA-GC1; Advanced Gastric Carcinoma; treatment response
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Detection of levels of circulating EV-derived lncRNA-GC1 — For patients with gastric cancer receiving neo-adjuvant chemotherapy, the dynamic changes of EV-derived lncRNA-GC1 was detected to identify whether is can serve as a monitoring biomarker for treatment response.

SUMMARY:
The investigators hope that through the analysis and research to find determine whether lncRNA-GC1 could serve as a non-invasive biomarker for monitoring the neo-adjuvant chemotherapy response for personalized medicine for gastric cancer.

DETAILED DESCRIPTION:
The LncRNA-GC1could noninvasively track dynamics of tumor burden and has been proposed as a real-time biomarker that can provide both predictive and prognostic values. But the value in monitoring the neo-adjuvant chemotherapy response is unclear. The investigators hope that through the analysis and research to find determine whether lncRNA-GC1 could serve as a monitoring biomarker for patients with gastric cancer receiving neo-adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age≥ 18 years old
* Histologically confirmed gastric adenocarcinoma
* radiographically identified as advanced gastric cancer

Exclusion Criteria:

* Other previous malignancy within 5 year
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study
* Pregnancy or lactation period
* Legal incapacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample Shanxi - Hospital and community sample Beijing -Hospital
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Detection of levels of circulating exosomal lncRNA-GC1 | Through study completion, an average of 1 year
  Levels of circulating exosomal lncRNA-GC1 are detected by RT-PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital Ethics Committee, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data may be shared until the final results published.